CLINICAL TRIAL: NCT04843527
Title: Evaluation of Flash Continuous Glucose Monitoring to Reduce Hyperglycemia in People
Brief Title: Evaluation of Flash Continuous Glucose Monitoring to Reduce Hyperglycemia in People With T2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ADC-US-RES-19185
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- FreeStyle Libre (Active Comparator): Subjects will be randomized to use the FreeStyle Libre Flash Glucose Monitoring System to manage their diabetes.
  Interventions: Device: FreeStyle Libre System
- FreeStyle Libre plus food logging (Active Comparator): Subjects will be randomized to use the FreeStyle Libre Flash Glucose Monitoring System and a food logging smartphone application to manage their diabetes.
  Interventions: Device: FreeStyle Libre System plus food app

INTERVENTIONS:
Device: FreeStyle Libre System — FreeStyle Libre Flash Glucose Monitoring System
  Arms: FreeStyle Libre
Device: FreeStyle Libre System plus food app — FreeStyle Libre Flash Glucose Monitoring System and Smartphone Food Logging application
  Arms: FreeStyle Libre plus food logging

SUMMARY:
A multi-center, randomized, prospective, non-significant risk study to compare the impact of the FreeStyle Libre Flash Glucose Monitoring System with and without a food logging smartphone application on reducing time above 180 mg/dL in subjects with type 2 diabetes who are not adequately controlled on their existing oral anti-diabetes medication regimen.

DETAILED DESCRIPTION:
Approximately 350 subjects will be enrolled to obtain at least 84 randomized subjects,approximately 42 subjects per arm. Subjects will be randomized to use either the FreeStyle Libre Flash Glucose Monitoring System or FreeStyle Libre Flash Glucose Monitoring System with a food logging smartphone application to manage their diabetes.

The subsequent impact on reducing the amount of time spent above 180 mg/dL will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject has been diagnosed with type 2 diabetes.
* HbA1c greater than or equal to 7.5% and less than or equal to 12%
* Subject is on at least 1 diabetes medication in the classes of metformin, SGLT-2 inhibitors, GLP-1 agonists and DPP-4 inhibitors.
* Subject owns a compatible smartphone
* Subject agrees to a 3-month period of no diabetes medication changes.
* Subject is willing to make diet and lifestyle changes in response to education and glucose data

Exclusion Criteria:

* Subject is currently on insulin therapy or sulfonylurea-based medications.
* Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
* Subject is known to be pregnant at the time of study enrollment (applicable to female subjects only).
* Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Impact on time above 180 mg/dL | Three (3) months
  To assess the impact of the FreeStyle Libre Flash Glucose Monitoring System with and with food logging app on time above 180 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care Inc
Locations (4):
- United States (4):
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - HealthPartners Institute dba International Diabetes Center, Minneapolis, Minnesota
  - UMPC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No